CLINICAL TRIAL: NCT07089069
Title: Intensity-Dependent Effects of 4-week Transcranial Direct Current Stimulation on Motor Learning in Healthy Young Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Sport University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025044H
Record Dates: First submitted 2025-07-20; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Transcranial Direct Current Stimulation (tDCS)
Keywords: Transcranial Direct Current Stimulation; motor learning; Healthy young adults

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1 mA transcranial direct current stimulation (Experimental): The participants will receive 1 mA transcranial direct current stimulation (tDCS) over primary motor cortex(M1) intervention for a period of four weeks (10 sessions), but the participants will be blinded of what kind of intervention they are receiving.
  Interventions: Device: 1 mA transcranial direct current stimulation
- 2 mA transcranial direct current stimulation group (Experimental): The participants will receive 2 mA transcranial direct current stimulation (tDCS) over primary motor cortex(M1) intervention for a period of four weeks (10 sessions), but the participants will be blinded of what kind of intervention they are receiving.
  Interventions: Device: 2 mA transcranial direct current stimulation
- 3 mA transcranial direct current stimulation group (Experimental): The participants will receive 3 mA transcranial direct current stimulation (tDCS) over primary motor cortex(M1) intervention for a period of four weeks (10 sessions), but the participants will be blinded of what kind of intervention they are receiving.
  Interventions: Device: 3 mA transcranial direct current stimulation
- sham transcranial direct current stimulation group (Sham Comparator): The participants will receive sham transcranial direct current stimulation (tDCS) over primary motor cortex(M1) intervention for a period of four weeks (10 sessions), but the participants will be blinded of what kind of intervention they are receiving.
  Interventions: Device: sham transcranial direct current stimulation

INTERVENTIONS:
Device: 3 mA transcranial direct current stimulation — The intervention will be conducted using a battery-powered stimulator (TCS-E2000, Shenzhen Yingchi Technology Co., Ltd) through a pair of saline-soaked sponge electrodes (5 cm × 7 cm).The stimulation intensity will be set at 3 mA. The stimulation will last for 20 minutes each time, with a 10 s fade-in period at the start and a 10-s fade-out period at the end of stimulation. The participants will receive intervention lasting for four weeks(10 sessions).The anodal electrode will be placed over the primary motor cortex (M1), and the reference electrode will be positioned at the center of the forehead.
  Arms: 3 mA transcranial direct current stimulation group
Device: 2 mA transcranial direct current stimulation — The intervention will be conducted using a battery-powered stimulator (TCS-E2000, Shenzhen Yingchi Technology Co., Ltd) through a pair of saline-soaked sponge electrodes (5 cm × 7 cm).The stimulation intensity will be set at 2 mA. The stimulation will last for 20 minutes each time, with a 10 s fade-in period at the start and a 10-s fade-out period at the end of stimulation. The participants will receive intervention lasting for four weeks(10 sessions).The anodal electrode will be placed over the primary motor cortex (M1), and the reference electrode will be positioned at the center of the forehead.
  Arms: 2 mA transcranial direct current stimulation group
Device: 1 mA transcranial direct current stimulation — The intervention will be conducted using a battery-powered stimulator (TCS-E2000, Shenzhen Yingchi Technology Co., Ltd) through a pair of saline-soaked sponge electrodes (5 cm × 7 cm).The stimulation intensity will be set at 1 mA. The stimulation will last for 20 minutes each time, with a 10 s fade-in period at the start and a 10-s fade-out period at the end of stimulation. The participants will receive intervention lasting for four weeks(10 sessions).The anodal electrode will be placed over the primary motor cortex (M1), and the reference electrode will be positioned at the center of the forehead.
  Arms: 1 mA transcranial direct current stimulation
Device: sham transcranial direct current stimulation — The intervention will be conducted using a battery-powered stimulator (TCS-E2000, Shenzhen Yingchi Technology Co., Ltd) through a pair of saline-soaked sponge electrodes (5 cm × 7 cm).The intervention will last for 20 minutes each time, with a 10 s fade-in period at the start and a 10-s fade-out period at the end of stimulation，but there is not current in between. The participants will receive intervention lasting for four weeks(10 sessions).The anodal electrode will be placed over the primary motor cortex (M1), and the reference electrode will be positioned at the center of the forehead.
  Arms: sham transcranial direct current stimulation group

SUMMARY:
The goal of this clinical trial is to investigate the effects of different intensities of transcranial direct current stimulationover primary motor cortex on motor learning in healthy adults. The main question it aims to answer is:

Which intensity of tDCS can best improve motor learning? Researchers will compare 1 mA, 2 mA, and 3 mA tDCS to sham tDCS to see which intensity of tDCS is most effective in improving the ability of motor learning.

Participants will be randomly divided into four groups and receive 4 different intensities of tDCS(1 mA, 2 mA, 3 mA and sham tDCS),and will be blinded to the type of tDCS they received. We hypothesized that anodal tDCS at 2 mA would produce the most substantial improvement in motor learning.

DETAILED DESCRIPTION:
The present study aimed to investigate the effects of different intensities of tDCS-specifically 1 mA, 2 mA, and 3 mA-on motor learning in healthy adults. Both the acute effects following a single tDCS session and the cumulative effects after a 4-week intervention (10 sessions) were evaluated. Additionally, the study aimed to determine whether improvements in motor learning induced by 4 weeks of repeated tDCS would be sustained one week after completion of the intervention. We hypothesized that anodal tDCS at 2 mA would produce the most substantial improvement in motor sequence learning, both following a single session and after a 4-week intervention, compared to 1 mA, 3 mA, and sham stimulation. Furthermore, we expected that the motor learning gains observed in the 2 mA group would be sustained one week post-intervention, indicating the persistence of tDCS-induced effects. In contrast, we anticipated minimal improvement in the 1 mA group due to insufficient stimulation intensity, and no additional or even reduced benefits in the 3 mA group compared to the 2 mA group.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 25 years; (2) normal or corrected-to-normal vision; (3) no history of pregnancy, cardiovascular disease, other physical impairments or illnesses, and no personal or family history of mental illness; (4) no implantation of any internal or external medical devices; and (5) right-handedness.

Exclusion Criteria:

-

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Sequence Reaction Time Task | Assessments will conducted before the intervention (Baseline), immediately after the first intervention (T1), at the end of 4 weeks (T2), and 1 week after the end of intervention (T3).
  In this task, a white circle appears above one of four horizontally arranged white squares on the computer screen with black background. Participans were instructed to press the proper button on the response pad (buttons H, J, K, L) using the corresponding finger of the right hand (index finger for button H, middle finger for button J, ring finger for button K, and small finger for button L) when the white circle appeared at the left side, middle-left side, middle-right side, or right side of the computer screen, respectively. Each session consists of eight blocks, with each block comprising 120 trials.

IPD SHARING:
Plan to Share IPD: Undecided
The specific contents of the IPD that can be shared have not yet been determined.